CLINICAL TRIAL: NCT03221764
Title: The Intra-Operative Application of Amiodarone Releasing Hydrogel to Prevent Postoperative Atrial Fibrillation in Patients Undergoing Lung Transplantation
Brief Title: Intraoperative Amiodarone to Prevent Atrial Fibrillation in Lung Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Victor Van Berkel, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16.1213
Record Dates: First submitted 2017-07-10; First posted 2017-07-19 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Atrial Fibrillation; Lung Transplant; Complications
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; CoSeal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Amiodarone with CoSeal administered with CO2 driver (Experimental): Lung Transplant Recipients who receive Intraoperative application of an Amiodarone containing hydrogel at the time of transplant.
  Interventions: Drug: Amiodarone with CoSeal; Device: CO2 driver

INTERVENTIONS:
Drug: Amiodarone with CoSeal — CoSeal Surgical Sealant (Baxter Healthcare) consist of 2 formulations of synthetic polyethylene glycols, a dilute hydrogen chloride solution along with a sodium phosphate/sodium carbonate solution. These separate solutions are mixed at the time of application to form a hydrogel. Amiodarone hydrochloride powder (1mg/kg) will be mixed with CoSeal at the time of application to form an amiodarone containing hydrogel. The dosing of amiodarone is based on previous study using amiodarone hydrogel in post-operative coronary artery bypass patients [8]. This hydrogel will be delivered utilizing a CO2 driver along the pulmonary vein and arterial anastomoses, and to the surface right and left atria.
  Other Names: Amiodarone with CoSealadministered with CO2 driver
Device: CO2 driver — The amiodarone hydrogel will be delivered utilizing a CO2 driver along the pulmonary vein and arterial anastomoses, and to the surface right and left atria.

SUMMARY:
This study will prospectively evaluate the use of an amiodarone releasing hydrogel applied to the pulmonary veins and atria at the time of lung transplantation. This study will include patients undergoing lung transplantation at Jewish Hospital, Louisville KY. The prospective group will be compared to historical controls from the same institution. Investigators will access medical records and database entries for those patients undergoing lung transplantation after January 1st 2005 in order to obtain matched controls for analysis. Informed consent will be obtained from the prospective cohort prior to patient enrollment. This pilot study will be used to obtain preliminary data in order to proceed with a larger randomized control trial.

DETAILED DESCRIPTION:
Approximately 1900 transplants are performed in the US annually. Lung transplantation remains the gold standard treatment for patients with end stage lung disease. This includes patients with range of etiologies such as Idiopathic Pulmonary Fibrosis, COPD and Cystic Fibrosis. One of the more common post-operative complications in patients undergoing lung transplantation is the development of atrial fibrillation. Recent studies have demonstrated that approximately 1/3 of patients will develop atrial fibrillation during their post-operative course. While it is uncertain if the development of post-operative atrial fibrillation affects survival, it does significantly increase length of hospital stay. Importantly, a portion of the patients that develop atrial fibrillation post-operatively will require cardioversion prior to discharge.

Currently one of the main stays of treatment for post-operative atrial fibrillation is systemic (oral or intravenous) amiodarone, which is a class III antiarrhythmic agent. While this particular drug is effective, it does carry the risk of several known complications. Due to the drug's pharmacokinetics, amiodarone concentrates in organs with high lipid content such as the thyroid, liver and lung. Amiodarone has several known adverse effects on the lung ranging from acute respiratory distress syndrome to more chronic disease such as Interstitial pulmonary fibrosis. Amiodarone can have detrimental effects on the liver which in rare cases could lead to cirrhosis. Additionally, amiodarone can cause thyrotoxicosis as early as a few weeks after the initiation of amiodarone.

The adverse events listed above are related to the cumulative dose of amiodarone. Typically, when amiodarone is initiated, patients receive a loading dose of 600-800mg daily until the cumulative dose reaches 10 grams, after which patients will receive 200mg daily as a maintenance dose. Minimizing the cumulative dose of amiodarone by using a local application, could mitigate the potential adverse drug toxicities. In a previous study, the application of an amiodarone releasing hydrogel performed intraoperatively was shown to significantly decrease the rates of post-operative atrial fibrillation in patients undergoing coronary artery bypass. Currently for patients undergoing lung transplantation, there is not a safe and effective measure available to prevent post-operative atrial fibrillation.

The Investigators aim to study the intraoperative application of an amiodarone containing hydrogel for prevention of post-operative atrial fibrillation in lung transplant patients.

In patients undergoing lung transplantation, post-operative atrial fibrillation is common and leads to prolonged hospital course and increased healthcare expenditures. Amiodarone is a main stay of therapy for atrial fibrillation, however this drug does have potential serious complications when administered systemically. The local application of amiodarone, could potentially decrease the rates of atrial fibrillation, while avoiding the systemic complications. This has the potential to decrease length of stay and decrease additional procedures (ie. Cardioversion) in patients undergoing lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative has signed Informed Consent Form (ICF)
* Undergoing lung transplant at the Jewish Hospital
* Age ≥ 18 years
* Subjects willing and able to comply with the follow up requirements of the study

Exclusion Criteria:

* Patients with previous history of atrial fibrillation.
* Patients with previously documented allergy or adverse reaction to amiodarone.
* Patients with previous ablation for atrial fibrillation
* Patients with an implantable pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor H van Berkel, MD, PHD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Patients undergoing who underwent application of an amiodarone containing hydrogel at the time of lung transplant.
Period: Overall Study
Arm/Group | Study Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.6 [60.3 to 70.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 4
Previous Coronary Artery Bypass [Count of Participants; unit: Participants] | 1
Previous Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 5
Diabetes [Count of Participants; unit: Participants] | 4
Hypertension [Count of Participants; unit: Participants] | 12
Cerebrovascular Disease [Count of Participants; unit: Participants] | 2
Smoking History [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Atrial Fibrillation
Description: Patient that developed atrial fibrillation after undergoing lung transplantation
Time Frame: Patients will be monitored for up to one year following lung transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 20
Participants | 6

2. Secondary Outcome: Atrial Fibrillation Requiring Intervention
Description: Patients that underwent cardioversion or ablation due to post operative atrial fibrillation
Time Frame: From transplant to discharge from hospital, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 20
Participants | 3

3. Secondary Outcome: Anti-Arrhythmic Medication at Discharge
Description: Patients that required anti-arrhythmic medication at the time of discharge for post operative atrial fibrillation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 20
Participants | 4

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=20)
Bradycardia (Cardiac disorders) | 0 (0) — Patients that developed post operative bradycardia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT03221764/Prot_SAP_ICF_001.pdf